CLINICAL TRIAL: NCT04398888
Title: Efficacy of a Modified Banxia Xiexin Decoction (BXD) for the "Wei-Pi" Syndrome (Postprandial Distress Syndrome): a Randomized, Waitlist Controlled Trial
Brief Title: Efficacy of a Modified Banxia Xiexin Decoction for the "Wei-Pi" Syndrome (Postprandial Distress Syndrome)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Buddhist Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-216
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2020-05

CONDITIONS: Postprandial Distress Syndrome
Keywords: Chinese medicine; Postprandial distress syndrome; Wei Pi; Banxia Xiexin Decoction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BXD treatment (Experimental): Participants will be diagnosed and treated by Chinese medicine practitioners (CMPs) with at least 5 years of clinical experience. CMPs will differentiate syndrome and prescript herbs in a semi-standardized protocol, which consists of a base Chinese medicine decoction, Banxia Xiexin Decoction (BXD), and the additional syndrome-specific herbs.
  The modified decoction will be prepared in a conventional decocting method at the Chinese medicine pharmacy in the clinic (HKBA-HKU CMCTR) and will be packaged into bags by the auto-decocting machines. Participants will take the decoction twice per day, 5 days per week, for 3 weeks.
  Interventions: Other: Banxie Xiexin Decoction (BXD)
- Waitlist (No Intervention): Participants in the waiting list control group will be observed for a three-week waiting period. Rescue medication is not restricted.

INTERVENTIONS:
Other: Banxie Xiexin Decoction (BXD) — A modified Banxie Xiexin Decoction based on Chinese medicine syndrome differentiation.
  Arms: BXD treatment

SUMMARY:
The study aims to evaluate the efficacy of a modified Banxia Xiexin Decoction (BXD) for Wei-Pi through a randomized, waitlist controlled trial.

DETAILED DESCRIPTION:
After being informed about the study plan, potential risk and benefits, all subjects will give written informed consent prior to participation and undergo eligibility screening. Eligible participants will be randomized, in a 1:1 ratio, into BXD group and waitlist group.

ELIGIBILITY:
Inclusion Criteria:

* Permanent resident of Hong Kong with age from 18 to 60
* Have a diagnosis of Wei-Pi (postprandial distress syndrome, ie. at least one of bothersome postprandial fullness (ie, severe enough to impact on usual activities) and bothersome early satiation (ie, severe enough to prevent finishing a regular-size meal) at least three days per week for the last three months, with symptom onset at least six months before diagnosis

Exclusion Criteria:

* Pregnancy or pregnancy planners
* Abnormal liver function (up to twofold the upper normal reference level of ALT)[14] or kidney function (estimated creatinine clearance < 80 mL/min)[15]
* History of diagnosed gastric structural abnormalities through endoscopy /History of gastric removal surgery
* Have G6PD deficiency
* Alcohol or drug abuser
* Taking Chinese medicine within one month
* Unable to read/understand and sign the informed consent document

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change of the Quality of Life Questionnaire for Functional Digestive Disorders | Change from baseline score at 3 weeks.
  Quality of Life Questionnaire for Functional Digestive Disorders (FDDQL)

SECONDARY OUTCOMES:
The Hospital Anxiety and Depression Scale | Weeks 0, 3, and 7
  The Hospital Anxiety and Depression Scale (HADS) consists of 14 items. Each item is scored from 0-3. Total score ranges between 0 and 21 for either anxiety or depression.
EQ-5D-5L | Weeks 0, 1, 2, 3, 4, and 7
  EuroQoL 5-dimension 5-level
Liver function test | Weeks 0 and 3.
  Serum Alanine transaminase (ALT) and Aspartate transaminase (AST).
Kidney function test | Weeks 0 and 3.
  Estimated Glomerular Filtration Rate (eGFR)
Quality of Life Questionnaire for Functional Digestive Disorders | Weeks 0, 3, and 7
  Quality of Life Questionnaire for Functional Digestive Disorders (FDDQL)

CONTACTS AND LOCATIONS:
Overall Officials: Haiyong CHEN, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong Buddhist Association - The University of Hong Kong Chinese Medicine Clinic cum Training and Research Centre (Wong Tai Sin District), Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sin SH, Wu J, Kang Y, Yip KHK, Kong NS, Wan H, Ng BFL, Chen H. Efficacy of modified Banxia Xiexin decoction in the management of Wei-Pi syndrome (postprandial distress syndrome): study protocol for a randomized, waitlist-controlled trial. Trials. 2021 Feb 12;22(1):135. doi: 10.1186/s13063-021-05078-y. PMID 33579349